CLINICAL TRIAL: NCT02387840
Title: Feasibility and Clinically Application of Magnetic Resonance Fingerprinting
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: technician left institution
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CASE7314; NCI-2015-00301 (Registry Identifier: CTRP)
Record Dates: First submitted 2015-02-27; First posted 2015-03-13 (Estimated); Results first posted 2021-01-12 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2020-12

CONDITIONS: Neurofibromatosis Type 1; Brain Tumor; Glioma
Keywords: Brain; Cancer; Neurofibromatosis type 1; NF1; Magnetic resonance fingerprinting; MRF
MeSH Terms: conditions — Neurofibromatosis 1; Brain Neoplasms; Glioma; Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (6):
- NF1-associated Optic Pathway Glioma (OPG) (Experimental): Patients with neurofibromatosis type 1 (NF1) associated OPG will be imaged by magnetic resonance imaging and magnetic resonance fingerprinting
  Interventions: Device: Magnetic Resonance Imaging; Device: Magnetic Resonance Fingerprinting
- NF1 without brain tumor (Experimental): Patients with NF1 without brain tumor will be imaged by magnetic resonance imaging and magnetic resonance fingerprinting
  Interventions: Device: Magnetic Resonance Imaging; Device: Magnetic Resonance Fingerprinting
- Without NF1 and with brain tumor exposed to therapy (Experimental): Patients without NF1 and with low grade gliomas exposed to therapy will be imaged by magnetic resonance imaging and magnetic resonance fingerprinting
  Interventions: Device: Magnetic Resonance Imaging; Device: Magnetic Resonance Fingerprinting
- Without NF1 and with untreated low grade brain tumors (Experimental): Patients without NF1 and with untreated low grade gliomas will be imaged by magnetic resonance imaging and magnetic resonance fingerprinting
  Interventions: Device: Magnetic Resonance Imaging; Device: Magnetic Resonance Fingerprinting
- Without NF1 and without brain tumors (Experimental): Patients without NF1 and without brain tumor will be imaged by magnetic resonance imaging and magnetic resonance fingerprinting
  Interventions: Device: Magnetic Resonance Imaging; Device: Magnetic Resonance Fingerprinting
- Brain tumors of assorted pathology (Experimental): Patients with brain tumors of assorted pathologies will be imaged by magnetic resonance imaging and magnetic resonance fingerprinting
  Interventions: Device: Magnetic Resonance Imaging; Device: Magnetic Resonance Fingerprinting

INTERVENTIONS:
Device: Magnetic Resonance Imaging — Patients will have a scan of soft tissue using magnetic field and radio frequency pulses.
  Other Names: MRI
Device: Magnetic Resonance Fingerprinting — Magnetic resonance fingerprinting (MRF) uses pseudo-randomized variation in acquisition parameters to generate a multi-parametric data signal that can be compared to signal patterns calculated from all possible combinations of parameters of interest. The closest match in signal patterns yields the parameters used to calculate the theoretical signal, in each voxel, and thus a map of all parameters of interest for that tissue. This process allows for rapid quantitation of MR relaxometry values (T1 and T2).
  Other Names: MRF

SUMMARY:
This study will look at the feasibility of using magnetic resonance fingerprinting (MRF) in children, adolescents and young adults (AYA) with and without brain tumors. This study will also look at subjects with and without neurofibromatosis type 1(NF1), a genetic disorder that affects the growth of nervous system cells. Further, it will explore potential ways of using of MRF signal measurements in children, adolescents, and young adults with brain tumors, including tissue characterization, looking at whether the treatment was effective, and finding metastasized tumors of unknown origin (occult tumors). To explore the feasibility and potential applications of MRF, this study will recruit up to 80 subjects but will stop once 10 subjects have usable data in each of six groups.

DETAILED DESCRIPTION:
Specific Aim 1: Demonstrate the feasibility of magnetic resonance fingerprinting (MRF) in children, adolescents and young adults (AYA) with and without brain tumors.

Specific Aim 2: Characterize the MRF signature of low-grade gliomas

Specific Aim 3: Determine whether MRF can identify occult tumor in subjects with low-grade glioma.

Specific Aim 4: Determine whether MRF can identify treatment effects in low-grade gliomas.

Specific Aim 5: Explore whether common brain tumors can be differentiated by comparing pre-operative MRF signature with pathologic diagnosis.

Outline: This study will examine the feasibility of MRF in children and AYA and determine whether quantitative measures of T1 and T2 relaxation times can be derived in subjects <35 years of age. Approximately 80 subjects will be evaluated and include subgroups where MRF may be of particular utility, including children and AYA subjects with brain tumors and subjects with neurofibromatosis type 1 (NF1). Additional aims will investigate the utility of MRF in these groups.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing MRI evaluation of the brain
* NF1 status will be determined by clinical exam or genetic testing
* NF1-associated Optic Pathway Glioma (OPG) will be defined as radiographic evidence of glioma along the optic nerve, chiasm, tract or radiation in a child with NF1
* Untreated low grade gliomas will be imaging-defined gliomas that have not yet been exposed to radiation or systemic chemotherapy. Those exposed to therapy will have had radiation and/or systemic chemotherapy more than 1 month prior to scans

Exclusion Criteria:

* History of mental retardation unrelated to brain tumor
* Presence of a genetic disorder other than NF1 that effects cognition or is associated with MR imaging abnormalities (e.g. tuberous sclerosis)
* History of cerebrovascular accident (stroke)
* Birth weight below five pounds, premature birth prior to 36 weeks of gestation, or ischemic episode at birth
* Major psychiatric diagnosis prior to neuro-oncological diagnosis

Max Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2015-03; Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah R Gold, MD, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Rainbow Babies and Children's Hospital, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Protocol enrollment was 35 but data are only available for 34 participants - Study team believes one participant's scan was never completed with MRF but because the study was terminated in 2018 with no further access to data this cannot be confirmed.
Period: Overall Study
Arm/Group | NF1-associated Optic Pathway Glioma (OPG) | NF1 Without Brain Tumor | Without NF1 and With Brain Tumor Exposed to Therapy | Without NF1 and With Untreated Low Grade Brain Tumors | Without NF1 and Without Brain Tumors | Brain Tumors of Assorted Pathology
Started | 4 | 6 | 6 | 8 | 4 | 6
Completed | 4 | 6 | 6 | 8 | 4 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants enrolled in study
Groups:
- Total: Total of all reporting groups
Arm/Group | NF1-associated Optic Pathway Glioma (OPG) | NF1 Without Brain Tumor | Without NF1 and With Brain Tumor Exposed to Therapy | Without NF1 and With Untreated Low Grade Brain Tumors | Without NF1 and Without Brain Tumors | Brain Tumors of Assorted Pathology | Total
Number analyzed (Participants) | 4 | 6 | 6 | 8 | 4 | 6 | 34
Age, Continuous [Median (Full Range); unit: Years] | 4.5 [2 to 22] | 17.5 [3 to 24] | 14 [10 to 21] | 15 [8 to 22] | 12.5 [0 to 20] | 14 [1 to 34] | 15 [0 to 34]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 4 | 6 | 3 | 0 | 18
  Male | 2 | 3 | 2 | 2 | 1 | 6 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 6 | 6 | 8 | 4 | 6 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 6 | 6 | 8 | 4 | 6 | 34
Region of Enrollment [Number; unit: participants]
  United States | 4 | 6 | 6 | 8 | 4 | 6 | 34

OUTCOME MEASURES:

1. Primary Outcome: Average Duration of MRF Sequence - Feasibility
Description: The duration of MRF sequence in minutes will be recorded as a measure of feasibility
Time Frame: Up to 1 year
Population: Participants enrolled in study
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | NF1-associated Optic Pathway Glioma (OPG) | NF1 Without Brain Tumor | Without NF1 and With Brain Tumor Exposed to Therapy | Without NF1 and With Untreated Low Grade Brain Tumors | Without NF1 and Without Brain Tumors | Brain Tumors of Assorted Pathology
Number analyzed (Participants) | 4 | 6 | 6 | 8 | 4 | 6
minutes | 11 (0) | 11 (0) | 11 (0) | 11 (0) | 11 (0) | 11 (0)

2. Secondary Outcome: Number of Patients With Evaluable T1 and T2 Relaxation Times on MRF Scans
Description: Number of patients which have evaluable scans at both T1 and T2
Time Frame: Up to 1 year
Population: Participants enrolled in study
Measure: Count of Participants; unit: Participants
Arm/Group | NF1-associated Optic Pathway Glioma (OPG) | NF1 Without Brain Tumor | Without NF1 and With Brain Tumor Exposed to Therapy | Without NF1 and With Untreated Low Grade Brain Tumors | Without NF1 and Without Brain Tumors | Brain Tumors of Assorted Pathology
Number analyzed (Participants) | 4 | 6 | 6 | 8 | 4 | 6
Participants | 4 | 6 | 6 | 8 | 4 | 6

3. Secondary Outcome: Comparison of Relaxometry MRI Scans Between Low Grade Gliomas and Healthy Brain Tissue
Description: Using Wilcoxon rank sum test to compare continuous variables, researchers will identify scans with significant difference in relaxometry between low-grade (composite of arms 1,3,4) and versus healthy brain tissue.
Time Frame: Up to 1 year
Population: Participants enrolled on arms 1,3 and 4. Combination of Arms 1, 3, and 4 for reporting was pre-specified in the study protocol. Each participant had a single tumor sample measured and a single normal-appearing white matter measured.
Measure: Mean (Standard Deviation); unit: milliseconds (ms)
Groups:
- Arms 1, 3, and 4 - Low Grade Gliomas: Arm 1: NF1-associated Optic Pathway Glioma (OPG) Arm 3: Without NF1 and with brain tumor exposed to therapy Arm 4: Without NF1 and with untreated low grade brain tumors
- Arms 1, 3, and 4 - Normal Appearing White Matter: Arms 1, 3, and 4 - Normal appearing white matter
Arm/Group | Arms 1, 3, and 4 - Low Grade Gliomas | Arms 1, 3, and 4 - Normal Appearing White Matter
Number analyzed (Participants) | 18 | 18
milliseconds (ms)
  T1 | 1355 (187) | 916 (78)
  T2 | 56 (19) | 38 (8)
Statistical Analysis 1: Comparison: Arms 1, 3, and 4 - Low Grade Gliomas vs Arms 1, 3, and 4 - Normal Appearing White Matter; Comparison of T1 values; Test type: Other — This test was a two-sample test using non-parametric data. A predefined margin was not used because no gold standard exists. A p-value of less than 0.05 was considered statistically different; p = 0.0002, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Arms 1, 3, and 4 - Low Grade Gliomas vs Arms 1, 3, and 4 - Normal Appearing White Matter; Comparison of T2 values; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.0003, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Combination of Relaxometry MRI Scans Between High Grade Gliomas and Healthy Brain Tissue
Description: Using Wilcoxon rank sum test to compare continuous variables, researchers will identify scans with significant difference in relaxometry between high-grade (arm 6) and versus healthy brain tissue.
Time Frame: Up to 1 year
Population: Participants in arm 6 had a measurable solid portion of HGG and were used for this analysis. Each participant had a single tumor sample measured and a single normal-appearing white matter measured.
Measure: Mean (Standard Deviation); unit: milliseconds (ms)
Groups:
- Arm 6 - High Grade Gliomas: Arm 6 - High Grade Gliomas
- Arm 6 - Normal Appearing White Matter: Arm 6 - Normal appearing white matter
Arm/Group | Arm 6 - High Grade Gliomas | Arm 6 - Normal Appearing White Matter
Number analyzed (Participants) | 3 | 3
milliseconds (ms)
  T1 | 1863 (70) | 979 (156)
  T2 | 91 (13) | 45 (7)
Statistical Analysis 1: Comparison: Arm 6 - High Grade Gliomas vs Arm 6 - Normal Appearing White Matter; Comparison of T1 values; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.081, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Arm 6 - High Grade Gliomas vs Arm 6 - Normal Appearing White Matter; Comparison of T2 values; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.081, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Comparison of Scans of Treated and Untreated Low Grade Gliomas (LGG)
Description: Using paired t-tests or non-parametric Wilcoxon signed rank tests, researchers will identify scans with significant differences in scans of treated and untreated tumors
Time Frame: Up to 1 year
Population: Participants enrolled in study. Combination of Arms for reporting was pre-specified in the study protocol
Measure: Mean (Standard Deviation); unit: milliseconds (ms)
Groups:
- Arms 1 & 4 - Untreated LGG: Arm 1: NF1-associated Optic Pathway Glioma (OPG) Arm 4: Without NF1 and with untreated low grade brain tumors
  The untreated LGG group consisted of Arm 4 and untreated participants from Arm 1.
- Arms 1 & 3 - Treated LGGs: Arm 1: NF1-associated Optic Pathway Glioma (OPG) Arm 3: Without NF1 and with brain tumor exposed to therapy
  The Treated LGG group consisted of Arm 3 and treated patients from Arm 1
Arm/Group | Arms 1 & 4 - Untreated LGG | Arms 1 & 3 - Treated LGGs
Number analyzed (Participants) | 9 | 7
milliseconds (ms)
  T1 | 1410 (180) | 1265 (181)
  T2 | 57 (15) | 47 (15)
Statistical Analysis 1: Comparison: Arms 1 & 4 - Untreated LGG vs Arms 1 & 3 - Treated LGGs; Comparison of T1 values; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.12, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Arms 1 & 4 - Untreated LGG vs Arms 1 & 3 - Treated LGGs; Comparison of T2 values; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.14, Wilcoxon (Mann-Whitney)

6. Other Pre Specified Outcome: Comparison of Relaxometry Values Between Tumors of Varying Pathology
Description: Descriptive statistics will be used to identify the T1 and T2 relaxation times for tumors of different types on pre-operative MRF scan
Time Frame: Up to 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 1 year
Arm/Group | NF1-associated Optic Pathway Glioma (OPG) | NF1 Without Brain Tumor | Without NF1 and With Brain Tumor Exposed to Therapy | Without NF1 and With Untreated Low Grade Brain Tumors | Without NF1 and Without Brain Tumors | Brain Tumors of Assorted Pathology
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/6 | 0/6 | 1/8 | 0/4 | 1/6
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/6 | 0/6 | 0/8 | 0/4 | 0/6
Other Adverse Events (participants affected / at risk) | 0/4 | 0/6 | 0/6 | 0/8 | 0/4 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-11-21): https://cdn.clinicaltrials.gov/large-docs/40/NCT02387840/Prot_SAP_000.pdf
  • Informed Consent Form (2017-10-26): https://cdn.clinicaltrials.gov/large-docs/40/NCT02387840/ICF_001.pdf